CLINICAL TRIAL: NCT03188198
Title: Phase II Randomized Study of R-CHOP V. Dose-Adjusted EPOCH-R in Untreated De Novo Diffuse Large B-Cell Lymphomas
Brief Title: Risk Adapted Therapy in Diffuse Large B Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mans lymphoma1
Record Dates: First submitted 2017-05-20; First posted 2017-06-15 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: Large B Cell Lymphoma
MeSH Terms: interventions — Rituximab; Etoposide; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A - R-CHOP (Active Comparator): Patients receive the following treatment:Rituximab 375 mg/m2 IV infusion on Day 1 prior to CHOP chemotherapy.Cyclophosphamide 750 mg/m^2 IV on Day 1.Doxorubicin 50 mg/m^2 IV on Day 1.Vincristine 1.4 mg/m^2 IV (2 mg cap) on Day 1.Prednisone 40 mg/m^2/day PO on Days 1-5.filgrastim or pegfilgrastim as defined in the protocol Required ancillary medications is administered during all cycles as defined in the protocol. Cycles will be repeated every 21 days for 6 treatment cycles. Restaging will occur after Cycles 4 and 6.
  Interventions:-Biological: rituximab-Drug: cyclophosphamide-Drug: doxorubicin-Drug: vincristine-Drug: prednisone-Drug: filgrastim-Drug: pegfilgrastim
  Interventions: Drug: rituximab, etoposide, cyclophosphamide, doxorubicin, vincristine,prednisone, filgrastim
- Arm B - DA-EPOCH-R (Experimental): Patients receive the following treatment: Cycle 1 Doses:Rituximab 375 mg/m^2 IV infusion on Day 1 prior to EPOCH chemotherapy. Doxorubicin 10 mg/m^2/day CIVI on Days 1-4.Etoposide 50 mg/m^2/day CIVI on Days 1-4. Vincristine 0.4 mg/m^2/day (no cap) CIVI on Days 1-4 (total 1.6 mg/m2 over 96 hours). Cyclophosphamide 750 mg/m^2 IV on Day 5 (following completion of 96 hour infusions). Prednisone 60 mg/m^2 PO BID on Days 1-5 Administer filgrastim 480 mcg subcutaneous daily from Day 6 until ANC > 5000 after the nadir (nadir usually between Days 10-12) Doses for subsequent cycles will be determined by the absolute neutrophil (ANC) or platelet nadir from the previous cycle. Cycles will be repeated every 21 days for a maximum of 6 cycles. Restaging will occur after Cycles 4 and 6.
  Interventions:
  -Biological: rituximab-Drug: cyclophosphamide-Drug: doxorubicin-Drug: vincristine-Drug: prednisone-Drug: etoposide-Drug: filgrastim
  Interventions: Drug: rituximab, etoposide, cyclophosphamide, doxorubicin, vincristine,prednisone, filgrastim

INTERVENTIONS:
Drug: rituximab, etoposide, cyclophosphamide, doxorubicin, vincristine,prednisone, filgrastim
  Other Names: rituximab:mabthera; etoposide:vepsid; cyclophosphamide:endoxan; doxorubcin:adriamycin

SUMMARY:
This randomized phase II trial is studying two different combination chemotherapy regimens to compare how well they work in treating patients with diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
objectives:

1. To compare the response rates and toxicity of R-CHOP versus DA-EPOCH-R in untreated CD20+ diffuse large B-cell lymphomas.
2. To compare the event-free survival of R-CHOP versus DA-EPOCH-R chemotherapy in untreated CD20+ diffuse large B-cell lymphomas.
3. To develop predictors of outcome of R-CHOP and DA-EPOCH-R chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically documented de novo CD20+ DLBCL with stage II, III or IV disease.

Stage I primary mediastinal (thymic) DLBCL is also eligible. Diagnosis should be based on an adequate tissue sample, including open biopsy or core needle biopsy.

Needle aspiration for primary diagnosis is unacceptable.

Patients must have one of the following WHO classification subtypes:

Diffuse large B-cell lymphoma (includes morphological variants: centroblastic, immunoblastic, T-cell/histiocyte rich, and anaplastic) Mediastinal (thymic) large B-cell lymphoma Intravascular large B-cell lymphoma Patients without adequate frozen material should have a biopsy performed to obtain material.

2. Patients may be entered if they have received prior limited field radiation therapy or a short course of glucocorticoids (< 10 days) for an urgent local disease complication at diagnosis (e.g., cord compression, SVC syndrome).

3. Age >16 years old. 4. ECOG Performance Status 0-2 5. If there is suspicion of cardiac disease, a cardiac ejection fraction must show LVEF > 45%.

6. Required Initial Laboratory Values (unless non-Hodgkin lymphoma):

* ANC ≥ 1000/μL
* Platelets ≥ 100,000/μL
* Creatinine≤ 1.5 mg/dL or creatinine clearance ≥ 50 cc/min
* Total Bilirubin ≤ 2 mg/dL (unless a history of Gilbert's Disease)

Exclusion Criteria:

* 1- Patients with an underlying low-grade lymphoma, such as a transformed lymphoma or low-grade lymphoma in the bone marrow, are not eligible.

  2- Patients with low international prognostic index are not eligible. 3- Prior cytotoxic chemotherapy or rituximab. Patients who have received chemotherapy for prior malignancies are not eligible.

  4- Active ischemic heart disease or congestive heart failure. 5- Known lymphomatous involvement of the CNS. A lumbar puncture prior to study is not required in the absence of neurological symptoms.

  6- Known HIV disease. Patients with a history of intravenous drug abuse or any other behavior associated with an increased risk of HIV infection should be tested for exposure to the HIV virus. Patients who test positive or who are known to be infected are not eligible.

  7- Pregnant and non-nursing. Treatment would expose an unborn child to significant risks. Women and men of reproductive potential should agree to use an effective form of contraception.

  8- Patients with active medical processes (e.g., uncontrolled bacterial or viral infection, bleeding) not related to their lymphoma should be excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Response rate | one year post-registration

SECONDARY OUTCOMES:
Event-free survival | Up to 3 years post-registration

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology center, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided